CLINICAL TRIAL: NCT06383858
Title: The Project of Gestational Hypertension and Preeclampsia Screening and Prevention
Brief Title: The Project of Gestational Hypertension and Preeclampsia Screening and Prevention Center
Status: Recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Dunjin Chen, Director of Guangzhou Institute of Obstetrics and Gynecology, The Third Affiliated Hospital of Guangzhou Medical University
Other Study IDs: [2024] Ethics Review NO.114
Record Dates: First submitted 2024-04-14; First posted 2024-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Preeclampsia; Maternal Deaths
Keywords: Preeclampsia; Placental growth factor (PlGF); Real-World Study; Screening; Prevention
MeSH Terms: conditions — Pre-Eclampsia; Maternal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All enrolled pregnant women will have 5 ml of peripheral blood drawn to detect PIGF levels when enrolling. Those with a high risk of preeclampsia need routine monitoring of PlGF or Soluble fms-Like Tyrosine Kinase 1（sFlt-1）/PlGF at 20-24+6 weeks and 30-30+6 weeks of pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Screening based on maternal factors: Pregnant women with low risk of pre-eclampsia assessment and no suspected pre-eclampsia symptoms in the later period are only followed up at delivery to register the outcome indicators. For pregnant women with high risk of preeclampsia evaluation, it is necessary to register the history of drug use (whether or not to use and the dosage), and follow up to register the outcome index at delivery.
  Interventions: Diagnostic Test: Screening method
- Screening based on FMF model: Preeclampsia risk assessment should be carried out at 11-13+6 weeks and 20-36+6 weeks of pregnancy. For low-risk pregnant women (PlGF≥100pg/ml or sFlt-1 /PlGF <38), it is suggested to closely monitor maternal blood pressure and conduct routine prenatal examination. The basic information of pregnant women, medical and obstetric history, physical examination information, ultrasonic examination data, serum markers (PlGF, sFlt-1) test results, pre-eclampsia risk assessment results, medication history and so on were registered in the study. For high-risk pregnant women (PlGF<100pg/ml or sFlt-1/PlGF ≥ 38), we should pay close attention to the changes of maternal blood pressure and proteinuria. Dynamic monitoring of PlGF or sFlt-1/PlGF should be carried out when necessary, and baseline information should also be registered after joining the group.
  Interventions: Diagnostic Test: Screening method

INTERVENTIONS:
Diagnostic Test: Screening method — All pregnant women in the group were screened for pre-eclampsia risk according to the clinical risk factors listed in NICE Guidelines (2019).
  Groups: Screening based on maternal factors
Diagnostic Test: Screening method — In the first trimester, pregnant women with routine MAP and PLGF (with UtA-PI detection conditions plus UtA-PI) were tested, and the risk of preeclampsia was evaluated based on Bayes rule combined with maternal factors. In the second and third trimester of pregnancy, routine determination of PLGF or sFlt-1/PLGF was used to evaluate the risk of preeclampsia.
  Groups: Screening based on FMF model

SUMMARY:
Preeclampsia is the main cause of illness and death in pregnant women and fetuses. Currently, there is no effective treatment for preeclampsia in clinical practice, and the fundamental treatment is still termination of pregnancy and placental delivery.

Therefore, early prediction of preeclampsia and targeted strengthening of high-risk pregnant women supervision, early intervention and diagnosis and treatment can greatly reduce the serious obstetric complications and perinatal maternal and fetal deaths caused by preeclampsia, which has significant social and clinical significance.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the influence of pre-eclampsia risk screening scheme based on maternal high-risk factors or pre-eclampsia risk assessment and management plan based on placental growth factor (PIGF) detection in the real medical world on the incidence of pre-eclampsia, maternal mortality and severe complications of pre-eclampsia, and to establish appropriate pre-eclampsia risk screening and prevention standards and guidelines for China population, so as to reduce the probability of maternal and fetal death and long-term chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1) Pregnant women who have been screened for pre-eclampsia risk according to the clinical risk factors listed in NICE guidelines (2019);
* 2) Based on the authoritative guideline of Figo and the consensus of experts in China, pregnant women who routinely use maternal factor +MAP＋PLGF±UtA-PI in the first trimester or PLGF or sFlt-1/PLGF in the second and third trimesters to assess the risk of preeclampsia.
* 3) Meet any of the above conditions, join the group voluntarily, and sign the informed consent form.

Exclusion Criteria:

* 1) Severe fetal malformation or abnormality (no fetal heartbeat);
* 2) Those who regularly use aspirin before joining the group;
* 3) There are obvious other abnormal signs, laboratory tests or other clinical d• iseases, which are judged by the researcher to be not suitable for participating in researchers;
* 4) Unable to obtain follow-up and delivery information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women ≥18 years old
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | 42 days after delivery
  The criteria for diagnosis and treatment of Hypertensive diseases in Pregnancy (2020) are implemented according to the Guidelines for Diagnosis and Treatment of Hypertensive Diseases in Pregnancy (2020), that is, systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after 20 weeks of pregnancy, accompanied by any one of the following: urinary protein quantity ≥0.3 g/24h, or urinary protein/creatinine ratio ≥0.3, or random urinary protein ≥ (+); No proteinuria, but accompanied by any of the following organs or systems: heart, lung, liver, kidney and other vital organs, or abnormal changes in the blood system, digestive system, nervous system, placenta - fetal involvement.

SECONDARY OUTCOMES:
Premature birth | <37 weeks
  Premature infants refer to all live births with a gestational age of<37 weeks
Fetal Growth Restriction | 42 days after delivery
  Affected by pathological factors such as maternal, fetal, and placental factors, fetal growth has not reached its expected genetic potential, often manifested as fetal ultrasound estimated weight or abdominal circumference being lower than the 10th percentile of the corresponding gestational age.
Severe complications of preeclampsia | 42 days after delivery
  When untreated, severe complications may occur in preeclampsia, such as eclampsia, liver rupture, stroke, pulmonary edema, or renal failure,

CONTACTS AND LOCATIONS:
Overall Officials: Dunjin Chen, Professor, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- FANG HE, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tang J, Xiao D, Yang S, Fang L, Liu H, Chen D, He F. sFlt-1/PlGF Ratio Predicts Short-Term Maternal-Fetal Outcomes in Chinese Hypertensive Pregnancies: A Prospective Cohort Study. Hypertension. 2026 Feb;83(2):e25022. doi: 10.1161/HYPERTENSIONAHA.125.25022. Epub 2025 Sep 15. PMID 40948128